CLINICAL TRIAL: NCT03229889
Title: Medication Facilitated Ureteral Access Sheath Deployment During Ureteroscopy and Endoscopic-Guided Percutaneous Nephrolithotomy: A Randomized Double-Blind Placebo Controlled Trial of Tadalafil, Tamsulosin and Combination
Brief Title: Trial of Tadalafil, Tamsulosin and Combination for Access Sheath Deployment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-3281
Record Dates: First submitted 2017-06-26; First posted 2017-07-26 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Nephrolithiasis
Keywords: Access Sheath; PCNL; Percutaneous Nephrolithotomy; Ureteroscopy; Alpha Blocker; Flomax; PDE-5 Inhibitor; Cialis; Phosphodiesterase Inhibitor
MeSH Terms: conditions — Nephrolithiasis | interventions — Tadalafil; Tablets; Tamsulosin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into 1 of 4 groups: Flomax + Placebo, Cialis + Placebo, Cialis + Flomax, Placebo + Placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both patients and treating surgeons (who are also on the study team) will be blinded. None physician researchers will be unblinded to tract and randomize patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Flomax + Placebo (Active Comparator): Patients will be prescribed Flomax 0.4Mg Capsule and given a bottle of placebo. They will be instructed to take 1 of each pill for the seven days prior to their surgery.
  Interventions: Drug: Flomax 0.4Mg Capsule
- Cialis + Placebo (Active Comparator): Patients will be prescribed Cialis 5Mg tablet and given a bottle of placebo. They will be instructed to take 1 of each pill for the seven days prior to their surgery.
  Interventions: Drug: Cialis 5Mg Tablet
- Cialis + Flomax (Active Comparator): Patients will be prescribed .4mg of Flomax and 5mg of Cialis. They will be instructed to take 1 of each pill for the seven days prior to their surgery.
  Interventions: Combination Product: Cialis + Flomax
- Placebo + Placebo (Placebo Comparator): Given 2 bottles of placebo. They will be instructed to take 1 of each pill for the seven days prior to their surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cialis 5Mg Tablet — Cialis is a PDE-5 inhibitor that has been shown to relax smooth muscle. Patients will be asked to 1 pill for 7 days prior to surgery.
  Other Names: Tadalafil
  Arms: Cialis + Placebo
Drug: Flomax 0.4Mg Capsule — Tamsulosin is an alpha-blocker that has been shown to relax smooth muscle in the genitourinary system. Patients will be asked to 1 pill for 7 days prior to surgery.
  Other Names: Tamsulosin
  Arms: Flomax + Placebo
Combination Product: Cialis + Flomax — Cialis is a PDE-5 inhibitor that has been shown to relax smooth muscle. Tamsulosin is an alpha-blocker that has been shown to relax smooth muscle in the genitourinary system. A combination of these two drugs may increase the relaxation effects in the ureter. Patients will be asked to 1 of each pill for 7 days prior to surgery.
  Other Names: Tamsulsoin; Tadalafil
  Arms: Cialis + Flomax
Drug: Placebo — This is plant cell based pill that contains no active ingredient. Patients will be asked to 1 pill for 7 days prior to surgery.
  Other Names: Inactive Drug
  Arms: Placebo + Placebo

SUMMARY:
Extensive literature exists on the use of alpha-blocker medications for the removal of kidney stones. Alpha blockers relax certain muscles and help small blood vessels remain open. They work by keeping the hormone norepinephrine (noradrenaline) from tightening the muscles in the walls of smaller arteries and veins, which causes the vessels to remain open and relaxed. This improves blood flow and lowers blood pressure. There are studies that demonstrate alpha-blockers decrease ureteral pressure and help the ureter "relax."

Recent studies have shown that phosphodiesterase inhibitors may also help with ureteral stone passing. A phosphodiesterase inhibitor is a drug that blocks an enzyme that inhibits relaxation of smooth muscle. This means that it can help smooth muscle, such as the muscle that lines the ureter, to relax. While ureteral relaxation is helpful in the passage of ureteral stones, our study seeks to use this finding by pretreating participants with an older generation alpha blocker or a phosphodiesterase inhibitor prior to passage of a ureteral access sheath in cases in which ureteroscopy is being used to approach a ureteral or renal stone.

By relaxing the ureter, it is possible that a larger access sheath can be safely placed. This may allow for facilitating passage of the ureteroscope and extraction of stone fragments while precluding the development of potentially damaging intrarenal pressure from the flow of irrigant. The ureteral access sheath also protects the ureter from damage during the procedure. Placement of the largest access sheath possible is helpful in that larger stone fragments can be retrieved, the flow of irrigant is improved, and the surgical field is kept clear of blood or debris. To date, nobody has studied whether use of an uro-selective alpha blocker, alone, or in combination with a 5 phosphodiesterase inhibitor will result in passage of larger access sheaths.

In this study participants will be randomized into 1 of 4 categories: Flomax (alpha-blocker), Cialis (5-phosphodiesterase inhibitor), a combination of the 2, or a placebo arm. In this study the placebo, or no active drug, is the current standard of care and will serve as a control from the other 3 groups.

DETAILED DESCRIPTION:
Technological improvements such as the miniaturization and development dual lumen ureteroscopes have improved the urologists' ability to treat urolithiasis1. The quality of flexible ureterorenoscopy is dependent on adequate visualization of the upper urinary tract. Adequate irrigation and visualization are compromised by debris from stone fragmentation and/or any bleeding during treatment. Fortunately, use of an ureteral access sheath (UAS) increases irrigant flow and reduces intrarenal pressure 2.

Ureteral access sheath technology was significantly improved by a member of our investigative team (RVC) thereby making it more widely acceptable3-5. The design changes allowed for easier deployment of the access sheath and the newer design was made to be kink resistant. This iteration of the device is easily deployed over a guidewire and has varying lengths such that it can be passed to the level of the stone in each case. Today's ureteral access sheaths range in size from 11-French to 16-French in diameter. The use of a ureteral access sheath has been shown to decrease intraoperative time, provide higher stone free rates, incur less cost due to shorter operating room times, and lead to fewer secondary procedures5,6. The access sheath should also, in theory, lower the risk of urinary tract infection due to decreased intrarenal pressure thereby resulting in less pyelovenous and less pyelolymphatic backflow. Lastly, use of an access sheath minimizes damage to the fragile flexible ureteroscope and thus increases their longevity while decreasing repair costs7.

Despite the above findings use of the UAS has not been universally embraced. A single study by Traxer et al., showed the incidence of low grade ureteric injury using UAS was 46% and that with serious injuries (i.e. urothelial tears) occurred in 13%8. However, a follow-up study by the same group showed no evidence of delayed long-term ureteral stricture formation; in fact, the patients who had a ureteral access sheath deployed there was a lower risk of post-operative complications9. Further, other studies have shown that the rate of ureteral stricture formation following use of a ureteral access sheath is 1.4% compared to a baseline rate of 1-3% during routine ureteroscopy without an access sheath10. In the afore cited study, the solitary occurrence of a post-ureteral access sheath ureteral stricture occurred at the ureteropelvic junction in a patient who underwent four endoscopic procedures for struvite stones; in all four surgeries, the access sheath was deployed at the level of iliac vessels well below the site of the patient's stricture10. Of note, porcine models have shown decrease ureteral blood flow following the acute deployment of a large access sheath, however over time the flow normalized and in follow-up there was no increase in post procedural ureteral stricture formation11.

Most urologists who place a ureteral access sheath do so without any pretreatment for ureteral relaxation. At our institution, the investigators routinely use alpha blockers (tamsulosin) as an adjunctive medical therapy to possibly relax the ureteral muscle; the medication is begun one week prior to surgery as it takes five days for the medicine to reach a steady state. It has been the investigator's experience that they are able to place larger ureteral access sheaths (i.e. 14 and 16 French size) with this approach. Additionally, examination of the ureter at the end of the procedure has shown minimal effect from placement of the access sheath; to date, the study team has not had any patient return with a post procedural ureteral stricture. Of note, it is the investigator's practice that if there is any resistance to deployment of the ureteral access sheath, then a smaller sized sheath is used; should the smaller sheath encounter resistance to its passage then a ureteral stent is placed and the procedure is postponed for a week. Stent placement in a ureter facilitates subsequent placement of an access sheath8,12.

An extensive literature exists on the role of alpha-blocker medications on the relaxation of ureteral smooth muscle13. This is due to the numerous alpha-1 receptors along the ureter, particularly in the distal ureter14,15. This knowledge originally led to the development of medical expulsive therapy in the treatment of ureteral stones. Several meta-analyses have shown that alpha blockers help passage of distal ureteral stones in the 5-10mm range, in less time and with less pain. The most extensively studied medication in this regard has been tamsulosin In addition to alpha blockade, recent in vitro studies have shown that phosphodiesterase-5 (PDE-5) inhibitors such as a tadalafil, commonly known by its tradename Cialis, also facilitate ureteral relaxation18-20. This has been substantiated by clinical studies which showed that sildenafil compared to placebo improved stone passage by 27%21. Further when tadalafil was added to tamsulosin the result was improved stone passage; the combined medications were well tolerated22,23.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing percutaneous nephrolithotomy (PCNL) or ureteroscopy (URS) for renal or proximal ureteral urolithiasis
* A documented sterile urine culture within 1-2 weeks of the procedure
* ≥ 18 years old
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

- Patients < 18-years-old

* Presence of ureteral stent or nephrostomy tube prior to scheduled procedure
* Patients requiring open, endoscopic, or laparoscopic procedure in the same setting as the intended URS or PCNL
* Planned concurrent bilateral endoscopic ureteral procedures
* Patients currently taking alpha-blockers within 14 days of surgery
* Patients taking PDE-5 inhibitors within 14 days of surgery
* Pregnant women
* Active urinary tract infection (UTI) or uncontrolled HIV
* Uncorrected coagulopathy
* Patients who cannot stop their blood thinners, and/or non-steroidal anti-inflammatory medications 5-7 days prior to the procedure
* Patients allergic to tamsulosin or tadalafil
* Patients with upcoming cataract surgery due to risk of floppy iris syndrome
* Patients with history of priapism
* Patients with hereditary retinitis pigmentosa
* Patients concurrently using nitrates for myocardial infarction (MI) or angina
* Patients with high risk cardiovascular disease: left ventricular outflow obstruction, MI in last 90 days, unstable angina, stroke in last 6 months, uncontrolled arrhythmias
* Patients with renal impairment (CrCl < 30 mL/min) or severe hepatic impairment (Child-Pugh score ≥ 10)
* Patients using CYP3A4 inhibitors such as clarithromycin, ritonavir, ketoconazole, or Iitraconazole

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-06-07 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Passage of 16F Access Sheath | This will be assessed immediately post-op per patient.
  Our primary objective is to assess the ability of a uroselective alpha-blocker (tamsulosin) and PDE-5 inhibitor (tadalafil), either alone or in combination will facilitate the passage of a 16F ureteral access sheath. Successful deployment will be defined as passage of the 16F ureteral access sheath into the proximal ureter or ureteropelvic junction. Difficulty in passing a 16F ureteral access sheath will be defined as a "failure". In this situation, we will place smaller ureteral access sheath (i.e. 11F or 14F), or opt to place a stent to dilate the ureter, and plan for surgery in the future; this is standard of care.

SECONDARY OUTCOMES:
Injury | This will be assessed immediately post-op per patient.
  Assessment of ureteral wall injury as defined by the post-ureteroscopic lesion score (PULS) as recorded during removal of the access sheath at the end of the surgical procedure
Complications | This will be assessed post-op per patient.
  Intraoperative complications will be recorded as defined by the Clavien-Dindo scale.
Adverse events | This will be assessed from the first day patients take the drugs until 1 weeks post-op.
  Incidence of adverse events with medications versus placebo as obtained during history on day of surgery, and during follow-up visit 1 week later
Stone-free status | This will be assessed immediately post-op as well as 3 months post-op.
  Stone free status as determined by low dose stone protocol CT scan per usual post-operative follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Landman, MD, Principal Investigator — UC Irvin Health
Locations (1):
- UC Irvine Health, Orange, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lusch A, Okhunov Z, del Junco M, Yoon R, Khanipour R, Menhadji A, Landman J. Comparison of optics and performance of single channel and a novel dual-channel fiberoptic ureteroscope. Urology. 2015 Jan;85(1):268-72. doi: 10.1016/j.urology.2014.09.032. PMID 25530400
- [Background] Landman J, Venkatesh R, Ragab M, Rehman J, Lee DI, Morrissey KG, Monga M, Sundaram CP. Comparison of intrarenal pressure and irrigant flow during percutaneous nephroscopy with an indwelling ureteral catheter, ureteral occlusion balloon, and ureteral access sheath. Urology. 2002 Oct;60(4):584-7. doi: 10.1016/s0090-4295(02)01861-7. PMID 12385911
- [Background] Takayasu H, Aso Y. Recent development for pyeloureteroscopy: guide tube method for its introduction into the ureter. J Urol. 1974 Aug;112(2):176-8. doi: 10.1016/s0022-5347(17)59675-5. No abstract available. PMID 4843325
- [Background] Monga M, Bhayani S, Landman J, Conradie M, Sundaram CP, Clayman RV. Ureteral access for upper urinary tract disease: the access sheath. J Endourol. 2001 Oct;15(8):831-4. doi: 10.1089/089277901753205843. PMID 11724124
- [Background] Kaplan AG, Lipkin ME, Scales CD Jr, Preminger GM. Use of ureteral access sheaths in ureteroscopy. Nat Rev Urol. 2016 Mar;13(3):135-40. doi: 10.1038/nrurol.2015.271. Epub 2015 Nov 24. PMID 26597613
- [Background] L'esperance JO, Ekeruo WO, Scales CD Jr, Marguet CG, Springhart WP, Maloney ME, Albala DM, Preminger GM. Effect of ureteral access sheath on stone-free rates in patients undergoing ureteroscopic management of renal calculi. Urology. 2005 Aug;66(2):252-5. doi: 10.1016/j.urology.2005.03.019. PMID 16040093
- [Background] Pietrow PK, Auge BK, Delvecchio FC, Silverstein AD, Weizer AZ, Albala DM, Preminger GM. Techniques to maximize flexible ureteroscope longevity. Urology. 2002 Nov;60(5):784-8. doi: 10.1016/s0090-4295(02)01948-9. PMID 12429296
- [Background] Traxer O, Thomas A. Prospective evaluation and classification of ureteral wall injuries resulting from insertion of a ureteral access sheath during retrograde intrarenal surgery. J Urol. 2013 Feb;189(2):580-4. doi: 10.1016/j.juro.2012.08.197. Epub 2012 Oct 8. PMID 22982421
- [Background] Traxer O, Wendt-Nordahl G, Sodha H, Rassweiler J, Meretyk S, Tefekli A, Coz F, de la Rosette JJ. Differences in renal stone treatment and outcomes for patients treated either with or without the support of a ureteral access sheath: The Clinical Research Office of the Endourological Society Ureteroscopy Global Study. World J Urol. 2015 Dec;33(12):2137-44. doi: 10.1007/s00345-015-1582-8. Epub 2015 May 14. PMID 25971204
- [Background] Delvecchio FC, Auge BK, Brizuela RM, Weizer AZ, Silverstein AD, Lallas CD, Pietrow PK, Albala DM, Preminger GM. Assessment of stricture formation with the ureteral access sheath. Urology. 2003 Mar;61(3):518-22; discussion 522. doi: 10.1016/s0090-4295(02)02433-0. PMID 12639636
- [Background] Lallas CD, Auge BK, Raj GV, Santa-Cruz R, Madden JF, Preminger GM. Laser Doppler flowmetric determination of ureteral blood flow after ureteral access sheath placement. J Endourol. 2002 Oct;16(8):583-90. doi: 10.1089/089277902320913288. PMID 12470467
- [Background] Miernik A, Wilhelm K, Ardelt PU, Adams F, Kuehhas FE, Schoenthaler M. Standardized flexible ureteroscopic technique to improve stone-free rates. Urology. 2012 Dec;80(6):1198-202. doi: 10.1016/j.urology.2012.08.042. PMID 23206763
- [Background] Hollingsworth JM, Rogers MA, Kaufman SR, Bradford TJ, Saint S, Wei JT, Hollenbeck BK. Medical therapy to facilitate urinary stone passage: a meta-analysis. Lancet. 2006 Sep 30;368(9542):1171-9. doi: 10.1016/S0140-6736(06)69474-9. PMID 17011944
- [Background] Edyvane KA, Trussell DC, Jonavicius J, Henwood A, Marshall VR. Presence and regional variation in peptide-containing nerves in the human ureter. J Auton Nerv Syst. 1992 Jun 15;39(2):127-37. doi: 10.1016/0165-1838(92)90053-j. PMID 1385511
- [Background] Itoh Y, Kojima Y, Yasui T, Tozawa K, Sasaki S, Kohri K. Examination of alpha 1 adrenoceptor subtypes in the human ureter. Int J Urol. 2007 Aug;14(8):749-53. doi: 10.1111/j.1442-2042.2007.01812.x. PMID 17681068
- [Background] Davenport K, Timoney AG, Keeley FX Jr. Effect of smooth muscle relaxant drugs on proximal human ureteric activity in vivo: a pilot study. Urol Res. 2007 Aug;35(4):207-13. doi: 10.1007/s00240-007-0100-x. Epub 2007 May 26. PMID 17530238
- [Background] Kobayashi S, Tomiyama Y, Hoyano Y, Yamazaki Y, Kusama H, Itoh Y, Kubota Y, Kohri K. Gene expressions and mechanical functions of alpha1-adrenoceptor subtypes in mouse ureter. World J Urol. 2009 Dec;27(6):775-80. doi: 10.1007/s00345-009-0396-y. PMID 19259685
- [Background] Taher A, Schulz-Knappe P, Meyer M, Truss M, Forssmann WG, Stief CG, Jonas U. Characterization of cyclic nucleotide phosphodiesterase isoenzymes in the human ureter and their functional role in vitro. World J Urol. 1994;12(5):286-91. doi: 10.1007/BF00191209. PMID 7866426
- [Background] Kuhn R, Uckert S, Stief CG, Truss MC, Lietz B, Bischoff E, Schramm M, Jonas U. Relaxation of human ureteral smooth muscle in vitro by modulation of cyclic nucleotide-dependent pathways. Urol Res. 2000 Apr;28(2):110-5. doi: 10.1007/s002400050147. PMID 10850633
- [Background] Gratzke C, Uckert S, Kedia G, Reich O, Schlenker B, Seitz M, Becker AJ, Stief CG. In vitro effects of PDE5 inhibitors sildenafil, vardenafil and tadalafil on isolated human ureteral smooth muscle: a basic research approach. Urol Res. 2007 Feb;35(1):49-54. doi: 10.1007/s00240-006-0073-1. Epub 2006 Nov 11. PMID 17102958
- [Background] Shokeir AA, Tharwat MA, Abolazm AE, Harraz A. Sildenafil citrate as a medical expulsive therapy for distal ureteric stones: A randomised double-blind placebo-controlled study. Arab J Urol. 2016 Mar;14(1):1-6. doi: 10.1016/j.aju.2015.12.001. Epub 2016 Jan 21. PMID 26966585
- [Background] Jayant K, Agrawal R, Agrawal S. Tamsulosin versus tamsulosin plus tadalafil as medical expulsive therapy for lower ureteric stones: a randomized controlled trial. Int J Urol. 2014 Oct;21(10):1012-5. doi: 10.1111/iju.12496. Epub 2014 Jun 3. PMID 24894533
- [Background] Kloner RA, Jackson G, Emmick JT, Mitchell MI, Bedding A, Warner MR, Pereira A. Interaction between the phosphodiesterase 5 inhibitor, tadalafil and 2 alpha-blockers, doxazosin and tamsulosin in healthy normotensive men. J Urol. 2004 Nov;172(5 Pt 1):1935-40. doi: 10.1097/01.ju.0000142687.75577.e4. PMID 15540759
- [Background] Schoenthaler M, Buchholz N, Farin E, Ather H, Bach C, Bach T, Denstedt JD, Fritsche HM, Grasso M, Hakenberg OW, Herwig R, Knoll T, Kuehhas FE, Liatsikos E, Liske P, Marberger M, Osther PJ, Santos JM, Sarica K, Seitz C, Straub M, Traxer O, Trinchieri A, Turney B, Miernik A. The Post-Ureteroscopic Lesion Scale (PULS): a multicenter video-based evaluation of inter-rater reliability. World J Urol. 2014 Aug;32(4):1033-40. doi: 10.1007/s00345-013-1185-1. Epub 2013 Oct 18. PMID 24135917